CLINICAL TRIAL: NCT07064070
Title: Technology-Based Resources to Increase Uptake of Sexual Health Services for Teens
Acronym: TRUST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-32013; U48DP006374 DP20-003: SIP20-00 (Other Grant/Funding Number: Center for Disease and Control); U48DP006374 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: mHealth Intervention
Keywords: mHealth; adolescent; sexual health; alone time; well child visit

STUDY DESIGN:
Intervention Model Description: participants have accessed to the intervention. Single arm study with pre and post design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participant will interact with four module on a secured website. (Experimental): The online modules included: General Communication, Talking about Relationships and Sexual Health, Parental Monitoring, and Check-up and Check-in (content focused on the importance of alone time). Modules were in English, Chinese, or Spanish
  Interventions: Behavioral: TRUST

INTERVENTIONS:
Behavioral: TRUST — The four online modules included: General Communication, Talking about Relationships and Sexual Health, Parental Monitoring, and Check-up and Check-in (content focused on the importance of alone time). Modules were in English, Chinese, or Spanish

SUMMARY:
Alone time with healthcare providers is vital for adolescents, as recommended by several professional organizations, as it enhances health service utilization, empowers adolescents to manage their health, and facilitates discussions on sensitive issues. Despite its importance, only 40% of adolescents have private conversations with clinicians during visits. mHealth technology offers a promising solution for effective interventions to promote alone time with providers for adolescents, parents, and healthcare providers. This pilot study aims to evaluate the preliminary efficacy of a technology-based intervention designed to increase alone time with providers during well-adolescent visits (WAVs) and its impact on trustworthiness, parent-adolescent communication, sexual risk communication, parental monitoring, and parental support. After providing consent, participants accessed a study website to complete a baseline survey, interact with four modules, and complete a post-test survey one month after WAVs. Surveys assessed alone time, trustworthiness, parent-adolescent communication, sexual risk communication, parental monitoring, and parental support.

DETAILED DESCRIPTION:
Background: Alone time with healthcare providers is critical for adolescents; several professional organizations recommend it. Alone time with providers promotes better utilization of health services, empowers adolescents to manage their health, and facilitates discussions on sensitive issues. However, only 40% of adolescents have private conversations with clinicians during visits. The advancement mHealth technology provides an excellent opportunity to deliver effective interventions to promote adolescent/provider alone time with adolescents, parents, and providers.

Objective: This pilot study aims to explore 1) the preliminary efficacy of a technology-based intervention designed to increase Alone time with providers during well-adolescent visits (WAVs) and 2) its impact on trustworthiness, parent-adolescent communication, sexual risk communication, parental monitoring, and parental support before and after the intervention.

Methods: A pre and post test design is utilized. After obtaining consent, participants accessed a study website to complete a baseline survey, interact with four modules, and complete a post-test survey one month after WAVs. Participants completed surveys assessing alone time, trustworthiness, parent-adolescent communication, sexual risk communication, parental monitoring, and parental support. Mixed model analysis and effect sizes for pre- and post-intervention outcomes were employed.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 11 and 17 years old
* The child can read and speak English
* The child has access to the internet (via phone or computer)
* The child has a well-child visit scheduled in the next 6 months.
* Mother could be included if they had an adolescent enrolled in this study
* Mother who speaks and reads English, Cantonese, Mandarin, or Spanish
* Mother has access to the internet.

Exclusion Criteria:

* Not have a well-child visit scheduled in the next 6 months.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Young Adult Health Care Survey (YAHCS) for Alone time | From enrollment to the end of intervention at 6 months
  Whether the adolescent had alone time with a healthcare provider (one-on-one communication without a parent) during the last well-adolescent visits (WAVs)

SECONDARY OUTCOMES:
Trustworthiness survey | From enrollment to the end of intervention at 6 months
  The construct of perceived trustworthiness was assessed using three items for adolescents and their mothers. Three items include: I can trust my mother/adolescent when we talk, b) my mother /adolescent keeps her promises to me, and c) my mother/adolescent is honest with me. Score ranges from 1 to 5, with a higher score indicating a higher level of trust.
Parent-Adolescent Communication Scale (PACS) | From enrollment to the end of intervention at 6 months
  A survey consists of 20 items that measure the quality of communication between adolescents and their parents. The score ranges from 1 to 5. Higher scores represent better parent-adolescent communication.
Parent-adolescent sexual risk communication scale (PTSRC-III): | From enrollment to the end of intervention at 6 months
  an 8-item scale used to assess the extent of sexual risk communication between adolescents and their parents. The scores range from 1 to 5 with a high score indicating a better parent-teen sexual risk communication. Higher values indicate more supportive parenting.
Supportive parenting survey | From enrollment to the end of intervention at 6 months
  Mothers reported how often they support their child (three items; 4-point Likert scale; Never to Always).

CONTACTS AND LOCATIONS:
Overall Officials: Jyu-Lin Chen, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Department of Family Health care Nursing, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JL, Raymond-Flesch M, Hoffmann TJ, Lin CX, Xu L, Koester KA. Evaluating the Preliminary Efficacy of the TRUST Intervention on Alone-Time and Communication During Well-Adolescent Visits: Quasi-Experimental Study. JMIR Pediatr Parent. 2025 Sep 8;8:e71433. doi: 10.2196/71433. PMID 40921058
- See also: TRUST Study — https://truststudy.ucsf.edu/

DOCUMENTS (1):
  • Informed Consent Form: Parent inform consent (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT07064070/ICF_000.pdf